CLINICAL TRIAL: NCT01484093
Title: Sequential Chemo-Radioimmunotherapy Followed by Autologous Transplantation for Patients With Untreated Advanced Stage Mantle Cell Lymphoma: A Phase I/II Trial
Brief Title: Sequential Chemo-Radioimmunotherapy Followed by Autologous Transplantation for Patients With Untreated Advanced Stage Mantle Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-095
Record Dates: First submitted 2011-11-29; First posted 2011-12-02 (Estimated); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Mantle Cell Lymphoma
Keywords: CYCLOPHOSPHAMIDE (CYTOXAN); CYTARABINE (ARA-C); DOXORUBICIN/ADRIAMYCIN; PREDNISONE; RITUXIMAB; TOSITUMOMAB (BEXXAR); Iodine; VINCRISTIN; Lymphoma; Chemo-Radioimmunotherapy; Autologous Transplantation; Untreated; 11-095
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma | interventions — tositumomab I-131

ARMS (1):
- R-CHOP-14R-HIDAC,followed by RIT/HDT/ASCR. (Experimental): This is a phase I/phase II multi-institution trial. The phase I part of the trial will determine the MTD of cytarabine. The phase II part of the trial will examine the efficacy of the proposed regimen by evaluating the 3-year event-free survival (EFS) in patients with untreated mantle cell lymphoma. All patients in the study in both phases will undergo induction and consolidation with R-CHOP 14R-HIDAC, followed by RIT/HDT/ASCR.
  Interventions: Other: R-CHOP-14R-HIDAC,followed by RIT/HDT/ASCR.

INTERVENTIONS:
Other: R-CHOP-14R-HIDAC,followed by RIT/HDT/ASCR. — INDUCTION: R-CHOP-14 CHEMOTHERAPY: 4 cycles every 2 weeks ± 1 day All patients in the study in both phases will undergo induction and consolidation with R-CHOP 14R-HIDAC, followed by RIT/HDT/ASCR. Patients will undergo restaging scans 12 to 14 days following completion of R-CHOP 14, with CT, and FDG-PET. Patients demonstrating at least a PR may proceed to consolidation with R-HIDAC. CONSOLIDATION: R- HIDAC CHEMOTHERAPY: 2 cycles every 3 weeks ± 2 days After R-HIDAC, restaging will occur 17-21 days post cycle 2 with CT scan (or FDG-PET, if this was positive following R-CHOP-14). Radioimmunotherapy Dosimetric dose is given approximately 4-5 weeks after completing cycle 2 of R-HIDAC. This is to be preferred 1 week post restaging scans 17-21 days post cycle 2 of RHIDAC, and up to 2 weeks post-scans will be acceptable only if required by 131 I Tositumomab availability.
  Other Names: HIGH DOSE CHEMOTHERAPY AND AUTOLOGOUS STEM CELL RESCUE (ASCR)Patients admitted to the hospital for high dose chemotherapy. The anticipated length of; stay is 3-4 weeks. 14 days ± 1 day following the administration of the therapeutic dose of Iodine 131 I; Tositumomab, patients will be admitted for high-dose chemotherapy. BEAM; will be administered

SUMMARY:
Mantle cell lymphoma (MCL) is a rare and aggressive type of lymphoma, with only about 3,000 cases diagnosed per year. MCL is considered a difficult cancer to treat. This study is being done to better understand how to treat MCL.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated advanced stage mantle cell lymphoma (Clinical stage 2 with abdominal involvement, stage 3 and stage 4).
* Histologic diagnosis confirmed by MSKCC pathologist as mantle cell lymphoma with Cyclin D1, or D2 and/or, D3 staining performed. Presence of measurable disease as determined by FDG-PET, CT, endoscopy, colonoscopy, or bone marrow biopsy.
* Ages 18-70.
* Transplant eligibility as confirmed by the Disease Management Team.
* KPS ≥ 70%.

Adequate organ function:

* WBC ANC ≥ 1000 cells/mcL and platelet count ≥ 100,000 cells/mcL unless felt to be secondary to underlying mantle cell lymphoma at which any count is permissible.
* Adequate renal function as determined by Cr < or = to 1.5 mg/dL or 24 hr creatinine clearance ≥ 50 ml/hr
* Adequate hepatic function as determined by total bilirubin < or = to 1.5x ULN (unless known Gilbert syndrome) and AST < or = to 5.0x ULN.
* Cardiac ejection fraction greater than or equal to 50% as determined by echocardiogram or MUGA.
* For patients ≥ age 60, a stress echocardiogram will be required, with same requirements as above.
* DLCO greater than or equal to 50% as determined by pulmonary function tests performed prior to initiation of treatment.
* Patients with positive Hepatitis B serologies will be treated per institutional guidelines.

Exclusion Criteria:

* Prior treatment for mantle cell lymphoma, including more than 7 days of steroids, immunotherapy, radioimmunotherapy, or chemotherapy. This does not include patients who have initiated R-CHOP at an outside institution within 2 weeks of enrollment.
* Patients using > or = to 10mg/day of steroids for any chronic medical condition
* Pregnant or breast-feeding. Note: Pre-menopausal patients must have a negative, serum HCG within 14 days of enrollment,.
* HIV positive or Hepatitis C antibody positive.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2011-11-29 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) | 1 year
  of HIDAC. For this study the MTD will be the dose at which no more than one grade 3 CNS toxic event (defined by CTCAE 4.0 as severe neurologic symptoms limiting self care ADLs') up to two weeks following HIDAC occurs among a 6 patient cohort. Phase I
3 year Event Free Survival (EFS) | 3 years
  from 67% (historical control) to 80 % in all patients. The EFS interval starts at enrollment date, and an event is defined as death from any cause or progression of disease. Patients who have completed the ASCT but elect to be removed from the study or lost to follow-up by the end of the third year will be counted as events as well. Phase II

SECONDARY OUTCOMES:
3-year Event Free Survival (EFS) | 3 years
  in subsets of patients with Ki-67 ≥ 30%
rates of complete remission (CR) | 1 year
  as defined by CT, FDG-PET and histology
Determine 3 year overall survival (OS). | 3 years
  Defined as last known follow up or date of death - date of diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Zelenetz, MD,PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan-Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- [Derived] Kumar A, Bantilan KS, Jacob AP, Park A, Schoninger SF, Sauter C, Ulaner GA, Casulo C, Faham M, Kong KA, Grewal RK, Gerecitano J, Hamilton A, Hamlin P, Matasar M, Moskowitz CH, Noy A, Palomba ML, Portlock CS, Younes A, Willis T, Zelenetz AD. Noninvasive Monitoring of Mantle Cell Lymphoma by Immunoglobulin Gene Next-Generation Sequencing in a Phase 2 Study of Sequential Chemoradioimmunotherapy Followed by Autologous Stem-Cell Rescue. Clin Lymphoma Myeloma Leuk. 2021 Apr;21(4):230-237.e12. doi: 10.1016/j.clml.2020.09.007. Epub 2021 Jan 1. PMID 33558202
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/